CLINICAL TRIAL: NCT04089761
Title: A Single Arm, Open Label, Multicenter Study of the Safety and Efficacy of Nerivio™ for the Acute Treatment of Migraine in Adolescents
Brief Title: Safety and Efficacy of Nerivio™ for the Acute Treatment of Migraine in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the outbreak of the COVID-19 pandemic in the USA on March 2020, all study sites stopped enrolling patients to the study
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCH004
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-06

CONDITIONS: Acute Migraine
Keywords: Migraine treatment, Adolescence

STUDY DESIGN:
Intervention Model Description: single arm, open-label, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active Device (Experimental): Treatment of acute migraine with an active form of Nerivio device
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — Nerivio™ is an FDA-authorized remote electrical neuromodulation (REN) device for the acute treatment of migraine with or without aura in patients 18 years old or above who do not have chronic migraine. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application.

SUMMARY:
Nerivio™ is an FDA-authorized remote electrical neuromodulation (REN) device for the acute treatment of migraine with or without aura in patients 18 years old or above who do not have chronic migraine. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism.

This is a prospective, single arm, open label, multicenter trial of the safety and efficacy of Nerivio™ for the acute treatment of migraine in adolescents

The study will be conducted in three phases:

Phase I - Run-in:

Phase II - Treatment phase:

Phase III (optional) - Free-use

DETAILED DESCRIPTION:
This open label study includes 3 phases and up to 4 visits. All visits will be conducted in the presence of a parent/guardian.

First visit - enrollment: The first visit will include screening, enrollment and training on the application in diary mode. The screening process will include an eligibility assessment and a urine pregnancy test. Following successful screening, enrollment interview and signing an informed consent by the parent/guardian and an informed assent by the participant. The participants will be trained to use the electronic diary application, installed on their own smartphones. The site personnel will be required to document the training session in the CRF. During this visit, participants will complete baseline questionnaires that included information on the frequency and severity of their migraine attacks, typical associated symptoms, use of preventive and acute treatments, and the effect that their migraine attacks have on their daily routine and quality of life.

Phase 1 - run-in phase: After the enrollment visit, participants will undergo a 4-week migraine diary phase aimed to collect baseline migraine characteristics and further assess eligibility. Participants will be asked to report in the application each migraine attack. These reports will be transferred by the application to the electronic data collection (EDC) system, where they will be collected and registered. Participants who did not have at least 3 migraine attacks will be excluded from the study. Eligibility will also be determined based on the compliance of participants to report the attacks within one hour from attack onset and report the pain level at 2 hours post-treatment in at least 66.7% of the reported attacks.

Second visit - Device training visit: Eligible participants who meet the run-in requirements will receive the Nerivio™ device. The device will be registered and connected by Bluetooth to their smartphone. During this visit, participants and their parent/guardian will be trained to use the device, including finding the optimal individual stimulation intensity level (perceptible but not painful). The site will also carefully review with the patient and parent/caregiver how to identify a qualifying migraine attack (see below) and provide detailed instructions on study procedures.

The individual intensity level identified during this visit will be recorded, and the participants will be asked to treat their migraine headaches with the device using the identified intensity. If the research staff recognizes that the participant cannot tolerate the feeling of the electrical stimulation, the participant may be withdrawn from the study.

Phase 2 -Treatment phase: Participants will be instructed to use the device for the treatment of 4 qualifying migraine attacks (see below) as soon as possible and always within 60 minutes of onset during a period of up to 8 weeks. Participants will be instructed to use the device with the intensity level identified during the device training visit (with a range of ±5 units) and make sure the stimulation is perceptible but not painful. Participants will be instructed to avoid taking rescue medications within 2 hours post-treatment. If medications are used, participants will be instructed to record in the app when and which medication was taken. The participants will use the app to record pain intensity levels (none, mild, moderate, or severe) at baseline, 2- and 24-hours post-treatment, and to record the presence/absence of associated migraine symptoms (nausea, photophobia, phonophobia) at baseline and 2 hours post-treatment. To assess functional disability, participants will also record at baseline, 2- and 24-hours post-treatment their response to the following question in their diary: "How do you rate your ability to do school-work or perform your usual activities?" using a 4-point scale ('as usual', 'some ability', 'a little ability', 'no ability at all'). At the beginning of each treatment, participants will also be asked to report the time elapsed from attack onset. Adverse events will be reported throughout this phase of the study.

Participants who do not achieve satisfactory relief at 2 hours post-treatment may treat again with the Nerivio™ device or may treat with usual care at that time or any time thereafter if the headache does not resolve. Participants will also be able to treat headache recurrence with the device. Attacks that are not treated with the device may be treated with usual care.

The first reported treatment will be considered a "training" treatment, aimed to verify that the participants use the device properly, and will only be included in the safety analysis. The efficacy evaluation will be performed on the first treatment of a qualifying attack (see below) following the training treatment (hereby termed "test treatment").

Third visit - Termination of the treatment phase and free-use phase initiation: Following the 8-week period of the treatment phase, participants will return to the clinic to return the device and fill questionnaires assessing satisfaction and user experience. All participants who complete the treatment phase will be offered to participate in an additional 8-week phase in which the device can be incorporate into usual care.

Phase 3 - Free-use phase: Participants will continue in an 8-week phase in which they will be able to use the device according to their preferences for the treatment of their migraine attacks.

Fourth (final) visit - End of study: Participants will return to the clinic following the end of the 8-week free-use phase, at which time they will return the device.

ELIGIBILITY:
Inclusion Criteria:

1. Participants age 12-17 years old at the time of informed consent, inclusive. 2. Participants have at least a 6-month history of headaches that meet the ICHD-3 diagnostic criteria for migraine with or without aura 3. History of at least 3 migraine attacks per month for each of the 2 months preceding study enrolment 4. Typical headache duration of at least 3 hours (when untreated or unsuccessfully treatment) 5. Stable migraine preventive medications during the 2 months prior to enrollment (no change in usage or dosage).

6. Participants have personal access to a smartphone (24/7) 7. Participants must be able and willing to comply with the protocol 8. Parents/Guardians must be able and willing to provide written informed consent 9. Participants must be able and willing to provide informed assent

Exclusion Criteria:

1. Participants with an implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker, cochlear implant).
2. Participants with congestive heart failure (CHF), severe cardiac or cerebrovascular disease.
3. Participants with epilepsy.
4. Medical use of cannabis or recreational use one month prior to enrollment.
5. Participants who have undergone nerve block (occipital or other) in the head or neck within the last 2 weeks
6. Treatment with onabotulinum toxin A (Botox) to the head and/or neck for 3 months before enrollment and/or during the study
7. Any history of anti-CGRP antibody treatment
8. Current participation in any other clinical study that includes treatment
9. Participants without basic cognitive and motor skills required for operating a smartphone.
10. Pregnant or breastfeeding females
11. Pure menstrual migraine
12. Participants who received parenteral treatments for migraine within the previous 2 weeks.
13. Participants with other significant pain, medical or psychological problems that in the opinion of the investigator may confound the study assessments
14. Participants who have previous experience with the device
15. Participants with arm circumference below 7.9 inches (20 cm)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hershey, MD, Principal Investigator — Director, Headache Center Cincinnati Children's Hospital Medical Center
Locations (12):
- United States (12):
  - Children's Hospital Colorado, Aurora, Colorado
  - Clinical Trials Solutions, Hialeah, Florida
  - Nicklaus children hospital, Miami, Florida
  - PANDA neurology, Atlanta, Georgia
  - Children Hospital New Orleans, New Orleans, Louisiana
  - Children Mercy Kansas City, Kansas City, Missouri
  - DENT neurology clinic, Amherst, New York
  - NYU Langone-Health, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Mercury Clinical Research, Houston, Texas
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hershey AD, Irwin S, Rabany L, Gruper Y, Ironi A, Harris D, Sharon R, McVige J. Comparison of Remote Electrical Neuromodulation and Standard-Care Medications for Acute Treatment of Migraine in Adolescents: A Post Hoc Analysis. Pain Med. 2022 Apr 8;23(4):815-820. doi: 10.1093/pm/pnab197. PMID 34185084

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study design
  Run-in:
  participants reported their migraine attacks, headache level and associated symptoms during a 4-weeks period.
  Treatment phase:
  Participants used the Nerivio device for the treatment of migraine attacks during a period of up to 8-week. participants reported their migraine attacks, headache level and associated symptoms.
  follow up (optional): Participants were asked to incorporate the Nerivio into their standard care according to their preferences.
Period: "Run In" Phase
Arm/Group | Active Device
Started | 60
Completed | 45
Not Completed | 15
Not completed — Not eligible to proceed to the treatment phase | 14
Not completed — Lost to Follow-up | 1
Period: "Treatment" Phase
Arm/Group | Active Device
Started | 45
Completed | 39
Not Completed | 6
Not completed — No evaluable data | 5
Not completed — Lost to Follow-up | 1
Period: "Follow Up" Phase (Optional)
Arm/Group | Active Device
Started | 27 (Due to the COVID-19 pandemic, Only 27 participants were able to continue to the "folllow Up" phase)
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Device
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 52
  More than one race | 0
  Unknown or Not Reported | 1
Average number of headache days per month [Mean (Standard Deviation); unit: Days per month] | 9.6 (4.6)
Migraine with aura [Count of Participants; unit: Participants] | 19
Triptan usage [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety of Nerivio Device
Description: Number of Participants with Device-Related Adverse Events
Time Frame: 12 weeks
Population: All subjects who entered to the treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 45
Participants | 1

2. Secondary Outcome: Pain Relief at 2 Hours Post Treatment
Description: The percentage of subjects reporting, for the test treatment, pain relief at 2 hours post-treatment without the use of rescue medication. Pain relief is defined as an improvement from severe or moderate pain to mild or no pain, or from mild pain to no pain. Pain level was reported using a 4-point Likert scale (0 -No pain, 1 - Mild pain, 2 - Moderate pain, 3- Severe pain)
Time Frame: 2 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 39
Participants | 28

3. Secondary Outcome: Pain-free at 2 Hours Post Treatment
Description: The percentage of subjects reporting, for the test treatment, no pain at 2 hours post-treatment without the use of rescue medication. Pain-free is defined as improvement from mild, moderate, or severe pain to no pain. Pain level was reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain, 3- Severe pain)
Time Frame: 2 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 39
Participants | 14

4. Secondary Outcome: Disappearance of Nausea at 2 Hours Post-treatment
Description: The percentage of subjects presented nausea at the baseline (T=0 hours) and reported disappearance of nausea at 2 hours post-treatment of the test treatment
Time Frame: 2 hours post treatment
Population: Only 22 subjects reported to have nausea at baseline (T=0 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 22
Participants | 12

5. Secondary Outcome: Disappearance of Photophobia at 2 Hours Post Treatment
Description: The percentage of subjects presented photophobia at baseline (T=0 hours) and reported disappearance of photophobia at 2 hours post-treatment of the test treatment
Time Frame: 2 hors post treatment
Population: Only 31 subjects reported to have photophobia at baseline (T=0 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 31
Participants | 13

6. Secondary Outcome: Disappearance of Phonophobia at 2 Hours Post Treatment
Description: The percentage of subjects presented phonophobia at baseline (T=0 hours) and reported disappearance of phonophobia at 2 hours post-treatment of the test treatment
Time Frame: 2 hours post treatment
Population: Only 25 subjects reported to have phonophobia at baseline (T=0 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 25
Participants | 10

7. Other Pre Specified Outcome: Sustained Pain Relief at 24 Hours Post Treatment
Description: The percentage of subjects achieving, for the test treatment, pain relief at 2 hours post-treatment without the use of rescue medication and no relapse of headache pain within 24 hours
Time Frame: 24 hours post treatment
Population: Only 22 of the 28 subjects with pain relief at T=2 hours reported their headache level at 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 22
Participants | 20

8. Other Pre Specified Outcome: Sustained Pain Free at 24 Hours Post Treatment
Description: The percentage of subjects achieving, for the test treatment, freedom from pain at 2 hours post-treatment without the use of rescue medication and no relapse of headache pain within 24 hours
Time Frame: 24 hours post treatment
Population: Only 11 of the 14 subjects with freedom from pain at T=2 hours reported their headache level at 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 11
Participants | 10

9. Other Pre Specified Outcome: Functional Disability at 2 Hours Post Treatment
Description: The percentage of subjects achieving improvement of at least one grade in functional disability in the test treatment at 2 hours post-treatment with no use of rescue medication
Time Frame: 2 hours post treatment
Population: Only 33 of the 35 subjects reported their functional disability score at both T=0 hours and T=2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 33
Participants | 23

10. Other Pre Specified Outcome: Functional Disability at 24 Hours Post Treatment
Description: The percentage of subjects achieving improvement of at least one grade in functional disability in the test treatment at 24 hours post-treatment with no use of rescue medication
Time Frame: 24 hours post treatment
Population: Only 29 of the 35 subjects reported their functional disability score at both T=0 hours and T=24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 29
Participants | 20

11. Post Hoc Outcome: Within-subject Consistency of the Pain Relief Response
Description: parcentage of subjects achieving pain relief at 2 hours in at least 50% of all their treatments
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 39
Participants | 26

12. Post Hoc Outcome: Within-subject Consistency of the Freedom From Pain Response
Description: percentage of subjects achieving freedom from pain at 2 hours in at least 50% of all their treatments
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device
Number analyzed (Participants) | 39
Participants | 13

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active Device
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 10/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Device (N=45)
Pain in the arm (Nervous system disorders) | 1 (1)
Common Cold (Reproductive system and breast disorders) | 1 (1)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Influenza (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Leg pain (General disorders) | 1 (1)
streptococcus pharyngitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Worsen migraine (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the outbreak of the COVID-19 pandemic in the USA, the enrollment of new patients was forced to be stopped.

An interim analysis was conducted at that point, to assess the statistical power of the data accumulated from the 60 patients enrolled which is approximately 50% of the planned sample size. Based on the results of this analysis, the data monitoring committee (DMC) determined that the study can be deemed completed for benefit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04089761/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04089761/ICF_001.pdf